CLINICAL TRIAL: NCT03801603
Title: Accelerating Uptake of the HPV Vaccine Among Rural and Native American Adolescents
Brief Title: Improving HPV Vaccination Rates Among Rural and Native American Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1330087
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: HPV Vaccinations
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPV Vaccination Training and Education (Experimental): Participants will be educated on the importance of HPV vaccination.
  Interventions: Behavioral: HPV vaccination training and education

INTERVENTIONS:
Behavioral: HPV vaccination training and education — 1) Training of providers and clinic staff on the importance of providing a strong HPV vaccination program and 2) HPV vaccination education for parents and the community.

SUMMARY:
This study will develop and implement a multi-level intervention aimed at improving human papillomavirus (HPV) vaccination rates at an Indian rural health clinic.

DETAILED DESCRIPTION:
The focus of this study is to develop, implement, and evaluate a human papillomavirus (HPV) vaccination program aimed at accelerating vaccine uptake among rural and Native American adolescents ages 11-17. HPV vaccination coverage with at least one dose remains disproportionately lower among rural adolescent compared to adolescents residing in urban areas and the rate of series completion is lower among Native American adolescent girls compared to non-Hispanic White adolescent girls.

ELIGIBILITY:
Inclusion Criteria:

* Clinic patients between the ages of 11-17 who are eligible for the HPV vaccine

Exclusion Criteria:

* None

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 263 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Clinic HPV Vaccination Rates | One year
  HPV vaccine uptake rates (initiation and completion of the 2-dose series) among clinic patients aged 11-17 as measured by the HPV ICD code from baseline to post.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis Comprehensive Cancer Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No